CLINICAL TRIAL: NCT06829316
Title: Epigenetic and Neurochemical Correlates of Bipolar Disorder: Investigating Key Biomarkers
Brief Title: Epigenetic and Neurochemical Correlates of Bipolar Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Salah Abdelhafeez Mostafa, Dr., Assiut University
Other Study IDs: Biomarkers in BD
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Disorder (BD)
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A 10 mL sample of venous blood will be collected from the antecubital vein under aseptic conditions and divided into two tubes. The first tube, containing anticoagulant (EDTA), will be centrifuged at 5000 rpm for 10 minutes. The separated plasma will then be stored at -20°C until biomarker analysis. The second tube will be stored as whole blood for subsequent DNA and RNA extraction.
  IL1B will be measured by DNA methylation of its gene using a DNA methylation kit (PCR).
  Serotonin receptors will be measured by their gene expression (PCR). Glutamic acid levels will be measured by ELISA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group I - Patients: Patients diagnosed with BD Diagnosis of BD will be established based on the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
- Group II: Unaffected first-degree relatives of patients with BD in group II
- Group III - Controls: Age and sex matched healthy individuals without a direct family history of BD as controls

SUMMARY:
Aim of Study:

* To assess DNA methylation of the IL1-B gene in individuals with BD compared to healthy controls.
* To evaluate the expression of 5-hydroxytryptamine (serotonin) receptors in BD and shed more light into its role into the pathophysioogy of BD.
* To measure differences of glutamic acid levels between study groups.
* To investigate correlations between these biomarkers among study groups, and their alignment with clinical presentations.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic and multifactorial psychiatric condition characterized by recurrent episodes of mania and depression, affecting approximately 2-3% of the global population. Despite extensive research, the precise pathophysiology of BD remains incompletely understood. Studies have shown that the pathophysiology of BD involves a combination of genetic, neurobiological, and environmental factors.

Classification of Bipolar Spectrum Disorders

They are generally divided into:

* BDI: This condition is characterized by alternating manic and depressive episodes.
* BDII: This condition is characterized by alternating depressive and hypomanic episodes.
* Cyclothymia: This condition is characterized by the alternation of mild depressive episodes and mild hypomanic episodes.
* BD not otherwise specified: in this condition, patients have symptoms of mania or hypomania that are too low or too brief to meet the diagnostic criteria for a syndrome.

Research on biomarkers for BD is ongoing, but no consensus has been reached on clinically diagnostic biomarkers. Recent findings also suggest that biomarkers may vary between early and late stages of BD. Neurochemical studies have shown that various neurotransmitters, such as serotonin, dopamine, glutamate (Glu) and GABA, may be involved in the pathophysiology of BD.

Epigenetics of BD: DNA Methylation of IL-1B (an Inflammatory Cytokine) Epigenetics involves hereditable reversible changes in gene function without altering the DNA sequence, such as DNA methylation, histone modification, and non-coding RNA regulation. While initially studied in normal development, epigenetic processes are now linked to various diseases including neurological and psychiatric disorders. These mechanisms reveal how gene-environment interactions contribute to the pathogenesis and comorbidity of such disorders.

DNA methylation is an epigenetic mechanism where a methyl group is added to the C5 position of cytosine, forming 5-methylcytosine. While gene expression in eukaryotes is regulated through various mechanisms, DNA methylation a common epigenetic tool used by cells to silence genes, effectively locking them in the "off" position.

IL 1B is a proinflammatory cytokine and has been implicated in the pathophysiology of BD. A meta-analysis revealed significantly higher peripheral IL-1β levels in patients with BD compared to controls, which supports inflammatory hypothesis of mood disorders.

Studies have found an inverse correlation between DNA methylation of the IL1B, IL6, and IL8 gene promoters and their corresponding mRNA levels, with this inverse correlation being most significant for IL1B.

Serotonin Receptors Serotonin (5-hydroxytryptamine, 5-HT) is a widely known monoamine neurotransmitter that regulates neural activity and various neuropsychological processes. Research on serotonin and its receptors continues to provide new biological insights with medical relevance across various organ systems. Serotonin plays a crucial role in regulating nearly all brain functions, and disruptions in the serotonergic system have been implicated in the pathogenesis of numerous psychiatric and neurological disorders.

The role of serotonin in the pathogenesis of mood disorders, particularly major (unipolar) depression, has been extensively studied, with most research indicating decreased central serotonergic function in major depressive disorder. However, the role of serotonin in the pathogenesis of BD has received comparatively less attention. The presence of manic episodes in BD suggests different or additional neurochemical abnormalities and highlights the need for studies of BD.

The serotonin 2A receptor (5-HT2A) is one of several subtypes of 5-HT receptors and has been implicated in mental disorders with complex and still poorly understood etiologies. It plays a role in cognitive processes, such as learning and memory, as well as neurogenesis.

Given the widespread distribution of this receptor in brain regions responsible for cognitive functions and social interaction, it is involved in disorders where these functions are impaired. Conditions such as schizophrenia, depression, obsessive-compulsive disorder (OCD), and attention-deficit hyperactivity disorder (ADHD) have been linked to alterations in the 5-HT2A receptor. Numerous drugs are designed to target this receptor.

Glutamate Glutamate is the primary excitatory neurotransmitter in the nervous system, with its pathways closely linked to those of other neurotransmitters. Glutamate receptors are present throughout the brain and spinal cord, in both neurons and glia. Dysfunction in glutamate signaling has significant effects in disease and injury.

Glutamate system dysfunction has been implicated in various mood disorders, with several studies highlighting reduced glutamate levels in certain brain regions of patients with major depressive disorder (MDD). In contrast, research on BD has yielded mixed results, with some studies showing altered glutamate activity while others report no significant changes.

ELIGIBILITY:
Inclusion Criteria:

* - Adults aged 18-45 with diagnosis of BD type I.
* Informed consent.

Exclusion Criteria:

* - Patients who have a concurrent severe illness or inflammatory disorders will be excluded. (e.g., other CNS disorders, autoimmune diseases, cancers... etc.)
* Current substance abuse.

Ages: 18 Months to 45 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A comprehensive medical history and physical examination will be conducted for all participants. Diagnosis of BD will be established based on the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker levels measurement | Within 6 months of sample collection
  Measurement and comparison of levels of DNA methylation of IL-1B gene, Serotonin receptor expression, and glutamic acid levels between study groups. Identifying correlations and possible ties to pathophysiology of BD.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahmood T, Silverstone T. Serotonin and bipolar disorder. J Affect Disord. 2001 Sep;66(1):1-11. doi: 10.1016/s0165-0327(00)00226-3. PMID 11532527
- [Background] Grezenko H, Ekhator C, Nwabugwu NU, Ganga H, Affaf M, Abdelaziz AM, Rehman A, Shehryar A, Abbasi FA, Bellegarde SB, Khaliq AS. Epigenetics in Neurological and Psychiatric Disorders: A Comprehensive Review of Current Understanding and Future Perspectives. Cureus. 2023 Aug 23;15(8):e43960. doi: 10.7759/cureus.43960. eCollection 2023 Aug. PMID 37622055
- [Background] Cherlyn SY, Woon PS, Liu JJ, Ong WY, Tsai GC, Sim K. Genetic association studies of glutamate, GABA and related genes in schizophrenia and bipolar disorder: a decade of advance. Neurosci Biobehav Rev. 2010 May;34(6):958-77. doi: 10.1016/j.neubiorev.2010.01.002. Epub 2010 Jan 7. PMID 20060416
- [Background] Kapczinski F, Dias VV, Kauer-Sant'Anna M, Brietzke E, Vazquez GH, Vieta E, Berk M. The potential use of biomarkers as an adjunctive tool for staging bipolar disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Nov 13;33(8):1366-71. doi: 10.1016/j.pnpbp.2009.07.027. Epub 2009 Aug 8. PMID 19666076
- [Background] Fortinguerra S, Sorrenti V, Giusti P, Zusso M, Buriani A. Pharmacogenomic Characterization in Bipolar Spectrum Disorders. Pharmaceutics. 2019 Dec 21;12(1):13. doi: 10.3390/pharmaceutics12010013. PMID 31877761
- [Background] Machado-Vieira R, Courtes AC, Zarate CA Jr, Henter ID, Manji HK. Non-canonical pathways in the pathophysiology and therapeutics of bipolar disorder. Front Neurosci. 2023 Aug 1;17:1228455. doi: 10.3389/fnins.2023.1228455. eCollection 2023. PMID 37592949